CLINICAL TRIAL: NCT05671796
Title: Phase 2, Double- Blind, Placebo- Controlled , Randomized Clinical Trial of Autologous Bone Marrow Stem Cell Transplantation in Patients With Subacute Spinal Cord Injury
Brief Title: Autologous Bone Marrow Stem Cell Transplantation in Patients With Subacute Spinal Cord Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SENAI CIMATEC (Other)
Collaborators: Oswaldo Cruz Foundation (Other); Federal University of Bahia (Other); Hospital Geral do Estado (Unknown); Hospital da Bahia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLC01/2021
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injury; Mesenchymal stem cells; Bone marrow
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell transplantation (Experimental): Two intrathecal autologous bone marrow stem cell transplantation of 1 ml solution containing 5x10,000,000 MSCs each with a 90-day interval between applications.
  Interventions: Genetic: Mesenchymal stem cell transplantation
- Placebo (Placebo Comparator): Two subcutaneous injections of 1 ml each, containing glycophysiological solution.with a 90-day interval between applications.
  Interventions: Other: Placebo

INTERVENTIONS:
Genetic: Mesenchymal stem cell transplantation — Patients will undergo two autologous bone marrow stem cell transplantation into the lesion area
  Arms: Mesenchymal stem cell transplantation
Other: Placebo — Patients will undergo two subcutaneous injections of 1 ml of glycophysiological solution into the lesion area by sham procedure
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of intrathecal administration of autologous mesenchymal stem cells in participants with subacute spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) constitutes a social and economic problem with the aggravating factor of being able to limit individual capacity, leading to a condition of unproductiveness and incapacity. At present, there is no effective treatment for recovering an injured spinal cord. Our research group was one of the pioneers in the study of mesenchymal stem cell therapies in the treatment of SCI, having carried out preclinical studies, as well as clinical studies with participants with complete spinal cord injuries, which demonstrated that stem cell transplantation mesenchymal (MSC) from autologous bone marrow was a safe and effective therapy in these studies. This project proposes the investigation of this therapy in participants with complete spinal cord injuries in the thoracolumbar region, in the subacute phase (defined between 3 to 6 months after the event), aiming to evaluate the safety and efficacy of the injection of mesenchymal stem cells. For this, we propose a double-blind, randomized clinical study to demonstrate the efficacy and safety of bone marrow MSC transplantation in participants with complete paraplegia, classified by ASIA Impairment Scale (AIS) grade A, by TRM, with subacute lesion. Forty participants will be referred by reference institutions and then recruited to be subsequently subjected to randomization, if eligible, with a group of 20 participants treated by intrathecal infusion of autologous MSCs, and another of 20 participants allocated to the control group, using a glucophysiological solution as a subcutaneous placebo. Each participant, after recruitment, will be monitored for a period of approximately 01 (one) year. The preparation of the CTMs will be done in accordance with the standards of good manufacturing practices. Both groups participating in the study will be submitted to pre- and post-treatment evaluations. The effectiveness of the therapy will be evaluated using the scale established by ASIA (American Spinal Injury Association) and the International Classification of Functioning, Disability and Health (ICF).

ELIGIBILITY:
Inclusion Criteria:

* Both sexes over 18 years old;
* Closed or open spinal cord injury at the thoracic or lumbar level in the subacute phase (between 3 and 6 months after the event);
* ASIA A rating.

Exclusion Criteria:

* Section of the spinal anatomy;
* Active infectious diseases;
* Terminal patients;
* Neurodegenerative diseases;
* Primary hematologic diseases;
* Bone reflecting increased risk for spinal puncture;
* Coagulopathies;
* Hepatic dysfunction;
* Pregnancy;
* Other medical complications that contraindicate surgery, including major respiratory complications;
* Participation in another clinical trial;
* Use of metal implants close to vascular structures (such as cardiac pacemaker or prosthesis) that contraindicate magnetic resonance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline ASIA scale and 12 Months after autologous mesenchymal stem cells transplantation in individuals with subacute spinal cord injury | Baseline and 12 months
  The International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), commonly referred to as the ASIA Exam, was developed by the American Spinal Injury Association (ASIA) as a universal classification tool for spinal cord injuries based on a standardized sensory and motor assessment.It involves both a Motor and Sensory examination to determine the Sensory Level and Motor Level for each side of the body (Right and Left), the single Neurological Level of Injury (NLI) and whether the injury is Complete or Incomplete. Elements of the scale include: Grade A: The impairment is complete, Grade B ,C and D: The impairment is incomplete with some differences between them.;Grade E: The patient's functions are normal

SECONDARY OUTCOMES:
Change from Baseline AIS scale and 12 Months after autologous mesenchymal stem cells transplantation | Baseline and 12 months
  American Spinal Injury Association Impairment Scale (AIS) is a standardized neurological examination used by the rehabilitation team to assess the sensory and motor levels which were affected by the spinal cord injury. The scale has five classification levels, ranging from complete loss of neural function in the affected area to completely normal. The results help the team set functional goals based on the neurological level of injury that is determined. Elements of the scale include: Grade A: The impairment is complete, Grade B ,C and D: The impairment is incomplete with some differences between them.;Grade E: The patient's functions are normal.
Improvement in quality of life, measured by the WhoQof-bref Questionnaire. | Baseline, 1 month, 6 months and 12 months
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale
Assessment of neuropathic pain by McGill Pain Questionnaire | Baseline, 1 month, 6 months and 12 months
  McGill Pain Questionnaire (MPQ) is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is a multi-dimesional tool for pain assessment and it has three components, which are the sensory intensity, the cognitive evaluation of pain and the emotional impact of pain.
Assessment sensory impairment after subacute spinal cord injury with von Frey filaments | Baseline, 1 month, 6 months and 12 months
  The mechanical sensitivity (Von Frey) test consists of thin calibrated plastic filaments that are applied to the plantar surface. Von Frey filaments of different gauges or stiffness are used to determine the threshold that elicits a hind paw withdrawal response. The mechanical withdrawal threshold is defined as the minimum gauge Von Frey filament that elicits a withdrawal reflex. The purpose of this test is to measure mechanical nociception in order to valuates the ability to detect a noxious stimulus.
Assessment sensory impairment after subacute spinal cord injury with Quantitative Sensory Test | Baseline, 1 month, 6 months and 12 months
  Quantitative sensory testing (QST) refers to psychophysical tests of sensory perception during the administration of stimuli with predetermined physical properties and following specific protocols. QST is able to capture and quantify stimulus-evoked negative and positive sensory phenomena,

CONTACTS AND LOCATIONS:
Overall Officials: Milena Soares, PhD, Study Director — SENAI CIMATEC; Augusto Mota, PhD, Principal Investigator — Hospital da Bahia
Locations (1):
- Senai Cimatec, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No